CLINICAL TRIAL: NCT05387733
Title: An Open-Label, Randomized Phase 2a Study to Evaluate the Efficacy and Safety of CBL-514 in Participants With Dercum's Disease Lipomas
Brief Title: A Study to Evaluate the Efficacy and Safety of CBL-514 in Participants With Dercum's Disease Lipomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Caliway Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBL-0201DD
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Dercum's Disease
Keywords: Adiposis Dolorosa; Lipedema; Lipomatosis; Skin Diseases; Lipid Metabolism Disorders; Metabolic Diseases; Connective Tissue Diseases
MeSH Terms: conditions — Adiposis Dolorosa; Lipedema; Lipomatosis; Skin Diseases; Lipid Metabolism Disorders; Metabolic Diseases; Connective Tissue Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CBL-514 Group 1 (Experimental): Eligible participants will be enrolled and randomized into one of 2 dose groups. Group 1 with 10 mg CBL-514 per injection.
  Interventions: Drug: 10 mg CBL-514 per injection
- CBL-514 Group 2 (Experimental): Eligible participants will be enrolled and randomized to one of 2 dose groups. Group 2 with 15 mg CBL-514 per injection.
  Interventions: Drug: 15 mg CBL-514 per injection

INTERVENTIONS:
Drug: 10 mg CBL-514 per injection — The total injection volume per lipoma will be based on the lipoma size, as determined by ultrasound. Dosing sceme is presented as below:
  Lipoma diameter of ≥1.0cm and ≤2.0cm - 1 injection (2 mL each); total of 10 mg CBL-514.
  Lipoma diameter of >2.0cm and ≤3.5cm - 2 injections (2 mL each); total of 20 mg CBL-514.
  Lipoma diameter of >3.5cm and ≤5.0cm - 3 injections (2 mL each); total of 30 mg CBL-514.
  Lipoma diameter of >5.0cm and ≤6.0cm - 5 injections (2 mL each); total of 50 mg CBL-514.
  Arms: CBL-514 Group 1
Drug: 15 mg CBL-514 per injection — The total injection volume per lipoma will be based on the lipoma size, as determined by ultrasound. Dosing sceme is presented as below:
  Lipoma diameter of ≥1.0cm and ≤2.0cm - 1 injection (3 mL each); total of 15 mg CBL-514.
  Lipoma diameter of >2.0cm and ≤3.5cm - 2 injections (3 mL each); total of 30 mg CBL-514.
  Lipoma diameter of >3.5cm and ≤5.0cm - 3 injections (3 mL each); total of 45 mg CBL-514.
  Lipoma diameter of >5.0cm and ≤6.0cm - 5 injections (3 mL each); total of 75 mg CBL-514.
  Arms: CBL-514 Group 2

SUMMARY:
This Phase 2 study will be an open-label and randomized study to assess the efficacy and safety of CBL-514 in participants with Dercum's Disease lipomas.

DETAILED DESCRIPTION:
This is a Phase 2a study to evaluate the efficacy and safety of CBL-514 injections in participants with Dercum's disease. It will employ an open-label, randomized study design.

Eligible participants will have at least 4 painful lipomas of appropriate size and up to 8 lipomas will be treated per subject. Eligible participants will be enrolled and randomized to 2 dose groups, with 6 participants per group. Each enrolled participant will receive up to 2 courses of their allocated dose of CBL-514 administered into selected lipomas, which the injection volume per lipoma will be based on the lipoma size, determined by ultrasound.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 years to 64 years old (at Screening), inclusive.
2. Body mass index (BMI) >18.5 kg/m2 at Screening and Day 1.
3. Has confirmed Dercum's disease and/or fulfills the following clinical criteria of Dercum's disease in localized nodular form. The final diagnosis of disease is in the opinion of the PI.

   1. Chronic pain (> 3 months) in the adipose tissue
   2. Pain in and around multiple lipomas.
4. Has at least 4 painful and well defined lipomas with a diameter of ≥1.0 cm and ≤6.0 cm as determined by ultrasound. Excluding lipomas in proximity to vulnerable anatomic structures, including the salivary glands, lymph nodes, muscles, and along the anatomic landmarks of the marginal mandibular nerve.
5. Generally considered healthy according to medical history, physical examination, electrocardiogram (ECG), and laboratory evaluation.
6. Voluntarily signs the Informed Consent Form (ICF) and, in the opinion of the PI or designee, is physically and mentally capable of participating in the study, and willing to adhere to study procedures.

Exclusion Criteria:

1. Women of childbearing potential (WOCBP) who are not willing to commit to an acceptable contraceptive regimen from the time of Screening and throughout study participation until 90 days after the last IP dose, or who are currently pregnant or lactating. Male participants who are not willing to commit to an acceptable contraceptive method. Female participants who are not WOCBP are not required to use contraception.
2. Participants that are unable to tolerate subcutaneous injections.
3. Participants that are diagnosed with another disorder with similar characteristics as Dercum's Disease.
4. Participants that are diagnosed with coagulation disorders or is receiving anticoagulant/antiplatelet therapy or medications or dietary supplements, which inhibit coagulation or platelet aggregation.
5. Participants who has fasting glucose concentration >200 mg/dL, delayed wound healing, bleeding risk, or any diabetic risks which, in the opinion of PI or designee, is inappropriate to participate in the study.
6. Participants with any clinically significant cardiac, hepatic, renal or neurologic/psychiatric disorders that in the opinion of the PI places the participant at significant risk.
7. Participants with positive blood screen for Hepatitis B surface antigen (HBsAg), Hepatitis C virus, or Human immunodeficiency virus (HIV).
8. Participants with clinical history of active primary or secondary immunodeficiency, autoimmune disease, or is undergoing chronic steroid or immunosuppressive therapy.
9. Participants with active, suspected, or prior history of malignancies within 5 years before Screening or being worked-up for a possible malignancy. Except adequately treated basal cell carcinoma of the skin and in situ squamous cell carcinoma of the skin would be eligible as per PI's discretion.
10. Participants with abnormal skin, local skin conditions, or body modifications at the treatment area, which in the opinion of the PI, is inappropriate for participation in the study, including but not limited to prior wound, scar tissue, infection in the treated area, or tatoo in the treated area.
11. Participants requiring continual use of the following therapeutic agents during the study: terfenadine, buspirone, fexofenadine, any medication that is known to strongly inhibit or induce CYP enzymes, sensitive CYP substrates or drugs with narrow therapeutic index, in the opinion of the Investigator, may affect the evaluation of the study product or place the participant at undue risk. If a participant requires the abovementioned therapeutic agents during the study for any reason, they should not be used for at least 2 days before dosing and until 1 day postdose.
12. Participants that undergone aesthetic procedure (eg, liposuction, cryolipolysis, ultrasonic lipolysis, low level laser therapy [LLLT], lipolysis injection) to the region to be treated before Screening or during the study.
13. Participants who are unable to receive local anesthesia.
14. Participants with known allergies or sensitivities to the IP or its components.
15. Participants that are in use of other investigational drug or device within 4 weeks prior to Screening.
16. Participant who has undergone vaccination (including with a live-attenuated vaccine) within 14 days prior to administration of the IP.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of CBL-514 following injection into lipomas or nodules of participants with Dercum's disease. | 0-84 days
  Evaluated the change of lipomas or nodules dimensions (as measured by ultrasound) after treatment with CBL-514 compared to Baseline.

SECONDARY OUTCOMES:
Efficacy of CBL-514 following injection into lipomas or nodules of participants with Dercum's disease. | 0-84 days
  Evaluated by percentage of lipomas or nodules with dimensions change and/or complete clearance (as measured by ultrasound) after treatment with CBL-514 compared to Baseline.
The change in pain of individual lipomas following CBL-514 injection in participants with Dercum's disease. | 0-84 days
  Assessed by change in pain assessment of individual lipomas evaluated by the Comparative Pain Scale compared to Baseline, where 0 is "no pain" and 10 is "worst pain".
The incidence of adverse events of special interests (AESI) as defined in the protocol. | 0-84 days
  Adverse events (AEs) will be assessed by recording of clinical responses (e.g. treatment-emergent adverse events (TEAEs), and injection site reactions (ISRs)).
The incidence of clinically significant abnormal findings as defined in the protocol. | 0-84 days
  Assessed by significant clinical changes in safety parameter (e.g. laboratory assessments, vital signs, ECGs, physical examinations).

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sheu, Study Director — Caliway Biopharmaceuticals Co., Ltd.
Locations (1):
- Karen L. Herbst, MD, PC, Tucson, Arizona, United States